CLINICAL TRIAL: NCT00007319
Title: Carotid Artery Intima-Media Thickness in HIV-Infected and Uninfected Adults: A Pilot Study
Brief Title: Carotid Artery Thickness in HIV Infected and Uninfected Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5078; AACTG A5078
Record Dates: First submitted 2000-12-16; First posted 2001-08-31 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2006-05

CONDITIONS: HIV Infections; HIV Seronegativity; Atherosclerosis
Keywords: HIV Protease Inhibitors; Risk Factors; HIV Seronegativity; Anti-HIV Agents; Carotid Artery; Tunica Intima; Atherosclerosis
MeSH Terms: conditions — HIV Infections; Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The intima-media thickness (IMT) test is a low cost, non-invasive way to measure the thickness of the carotid artery (the large artery in the neck). The purpose of this study is to compare the thickness of the carotid artery among HIV infected adults taking protease inhibitors (PIs), HIV infected adults not taking PIs, and HIV uninfected adults, and to examine how the thickness may change over time.

DETAILED DESCRIPTION:
Determination of clinical, lipid, and non-lipid risk factors has been the traditional approach for gauging an individual's risk for coronary artery disease (CAD). However, the IMT test, which uses sound waves to measure the thickness of the carotid artery, has been found to diagnose CAD and predict a person's risk for heart disease as well as or better than lipid and non-lipid risk factors. This study will use the IMT test to see if anti-HIV treatment and HIV infection affect a patient's risk of developing atherosclerosis (hardening of the arteries) by comparing carotid artery thickness among HIV infected adults taking PIs, HIV infected adults not taking PIs, and HIV uninfected adults.

There are 3 groups in this study. Group 1 will comprise HIV infected participants currently taking a PI-containing regimen. Group 2 will comprise HIV infected participants who are not taking PIs. Group 3 will comprise HIV uninfected participants. At each site, participants will be enrolled by "triads" consisting of an individual from each group. Each member of the triad will be closely matched by gender, age, smoking and menopausal status, race, and normal or hypertensive blood pressure. All 3 members of the triad must be identified before participants are registered to the study.

All participants will visit the clinic at Weeks 1, 24, 48, 72, 96, and 144 (3 years). At each visit, participants will have a physical exam, medical history and waist/hip ratio assessment, blood collection, and an IMT test. The absolute value for carotid IMT will be compared among the 3 groups. Viral load and CD4 counts will also be measured in Group 1 and 2 participants.

ELIGIBILITY:
Inclusion Criteria for Group 1

* HIV infected
* Have taken at least 1 PI continuously for 2 or more years and are currently taking at least 1 PI. Stopping therapy for 4 weeks or less for management of side effects or to change therapy is allowed.
* Viral load of 10,000 copies/ml or less

Inclusion Criteria for Group 2

* HIV infected
* Not currently receiving PIs or have not taken PIs in at least 3 months
* Not planning to initiate PI therapy in the few months following study entry
* Viral load of 10,000 copies/ml or less
* If not currently on anti-HIV treatment, must have been on treatment for at least 6 months in the past

Inclusion Criteria for Group 3

* HIV uninfected

Exclusion Criteria for All Groups

* Diabetes or current use of oral medications for diabetes
* Kidney disease
* ALT or AST greater than 2.5 times the upper limit of normal
* Hypothyroidism
* Family history (parents, brothers, sisters, or children) of heart attacks before age 55 in males and age 65 in females
* Alcohol or drug abuse
* Pregnant or plan to become pregnant during the study
* Body mass index (BMI) greater than 30
* Systemic chemotherapy or radiation therapy
* Systemic steroids (prednisone or equivalent) at doses greater than 5 mg/day for more than 30 consecutive days
* History of coronary heart disease or stroke (including chest pain, heart attack, or abnormal stress test)
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132

CONTACTS AND LOCATIONS:
Overall Officials: Judith S. Currier, MD, MSc, Study Chair — University of California, Los Angeles; Howard N. Hodis, MD, Study Chair — Atherosclerosis Research Unit, University of Southern California
Locations (10):
- United States (10):
  - Kaiser Foundation Hosp, Harbor City, California
  - Kaiser Permanente LAMC, Los Angeles, California
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of California, San Diego, San Diego, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Hawaii, Honolulu, Hawaii
  - Univ of Minnesota, Minneapolis, Minnesota
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Barbaro G. HIV infection, highly active antiretroviral therapy and the cardiovascular system. Cardiovasc Res. 2003 Oct 15;60(1):87-95. doi: 10.1016/s0008-6363(02)00828-3. PMID 14522410
- [Background] Calza L, Manfredi R, Chiodo F. Hyperlipidaemia in patients with HIV-1 infection receiving highly active antiretroviral therapy: epidemiology, pathogenesis, clinical course and management. Int J Antimicrob Agents. 2003 Aug;22(2):89-99. doi: 10.1016/s0924-8579(03)00115-8. PMID 12927947
- [Background] Mary-Krause M, Cotte L, Simon A, Partisani M, Costagliola D; Clinical Epidemiology Group from the French Hospital Database. Increased risk of myocardial infarction with duration of protease inhibitor therapy in HIV-infected men. AIDS. 2003 Nov 21;17(17):2479-86. doi: 10.1097/00002030-200311210-00010. PMID 14600519
- [Background] Penzak SR, Chuck SK. Management of protease inhibitor-associated hyperlipidemia. Am J Cardiovasc Drugs. 2002;2(2):91-106. doi: 10.2165/00129784-200202020-00003. PMID 14727985
- [Background] Varriale P, Saravi G, Hernandez E, Carbon F. Acute myocardial infarction in patients infected with human immunodeficiency virus. Am Heart J. 2004 Jan;147(1):55-9. doi: 10.1016/j.ahj.2003.07.007. PMID 14691419
- [Result] Currier JS, Kendall MA, Zackin R, Henry WK, Alston-Smith B, Torriani FJ, Schouten J, Mickelberg K, Li Y, Hodis HN; AACTG 5078 Study Team. Carotid artery intima-media thickness and HIV infection: traditional risk factors overshadow impact of protease inhibitor exposure. AIDS. 2005 Jun 10;19(9):927-33. doi: 10.1097/01.aids.0000171406.53737.f9. PMID 15905673